CLINICAL TRIAL: NCT04799860
Title: Act in Time- Implementation of Health Promotive Work-way in Primary Care Setting - Evaluation of Effect- and Implementation Process (AcTi)
Brief Title: Act in Time -Implementation of Health Promotive Work-way in Primary Care Setting (AcTi)
Acronym: AcTi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 275301
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: implementation; primary care; process evaluation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A pre-post-intervention design with control group will be used to evaluate intervention uptake and implementation process effectiveness from the perspective of managers, primary care professionals, patients, and organisation. Primary care settings in central Sweden will be supported in implementing a guideline-based health-promoting way of working including screening of life-style habits, measures taken according to evidence based recommendations and documentation. Strategies will include interactive education sessions, external and internal facilitators, audit and feedback, and tools from theories of leading change; tailored according to contextual and participant needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health promotive work-way (Experimental): Six primary care units that voluntarily enrolls as experimental units. The units will receive implementation support based on previous research and tailored to the specific prerequisits and context for each unit. Strategies includes involvement of target groups; informationa and interactive education;use of external and internal facilitators tarined for the purpose; systematic feedback and learning dialogs during the project. The implementation support will take approximately 12 months.
  Interventions: Behavioral: health promotive work-way
- Control (No Intervention): Six primary care centers of similar size and socioeconomic background in the population listed to each center.

INTERVENTIONS:
Behavioral: health promotive work-way — Clinical intervention: The patient is asked to fill in a screening form with life-style related questions. The caregiver takes adequate measures according to the recommendations of the national guideline and the filled in screeing form. The caregiver documents the measures taken.
  Implementation intervention as described previously: using tailored strategies to support implementation of the gudieline-based recommendations
  Arms: health promotive work-way

SUMMARY:
The study will support implementation of a health promotive work-way in primary care setting by using external and internal facilitators, with the aim to identify effective implementation strategies and to evaluate intervention uptake. Data will be collected from multiple perspecitves.

DETAILED DESCRIPTION:
Insufficient physical activity, hazardous use of alcohol, tobacco use and unhealthy eating habits increase the risk of cardiovascular diseases, cancer and type 2-diabetes. Health-promoting work reduces the disease risk and mortality and should thus be integrated in clinical care processes.

Despite support by the National guideline for prevention and treatment of unhealthy life-style habits, there is a chasm to bridge when integrating evidence into clinical practise. Prerequisites for changing work-ways are often underestimated and left to the individual co-workers to full fill on their own.

Too few patients are asked about life-style habits and too few receive evidence-based measures. The measures taken may also depend on sex, language, residence and caregiver's profession. The investigators strive to support the implementation of a health-promoting way of working that includes self-reporting of life-style habits before a visit and that takes measures for those with at least one unhealthy lifestyle habit.

The aim is to identify effective implementation strategies for health-promoting efforts in the primary care. The perceptions of barriers and opportunities when changing way of working from the target groups (leaders, co-workers, patients) will be used to enhance the possibility of successful implementation. Strategies are enhanced by theories of leading change. External and internal facilitators support the implementation.

The study will evaluate the effects and the implementation process at the level of leaders, patients, co-workers, facilitators and organisation in short (4-6 months) and long term (16-18 months).

The project provides generalizable knowledge on strategies to overcome the gap between evidence and praxis, contributing to utilize an existing synthesized knowledgebase regarding health-promoting and preventative workways in a Swedish primary care setting.

It is central for the health care system to identify successful implementation strategies in order to manage their future mission.

ELIGIBILITY:
Inclusion Criteria for co-workers:

* being a caregiver meeting patients and/or
* being assigned a role as internal or external facilitator in the project

Inclusion criteria for patients filling in the study specific questionnaire:

* 18 years or older
* visiting primary care units a specific time pre- or post implementation support

Inclusion criteria for personcentered processmapping:

* : having one or more unhealthy life-style habit 18 years or older

Inclusion criterina for managers:

* being a manager at a primary care unit or at higher level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change and trend from baseline documented codes in medical records | Change from baseline (6 months), through study completion up to 6 months after end of implementation support
  specific codes are used for measures related to the guideline recommendations for grade of advice for insufficient physical activity, unhealthy eating habits, hazardous use of alcohol and tobacco use and prescribed physical activity
Change and trend from baseline documented codes in medical records | Change from baseline (6 months), through study completion up to 18 months after end of implementation support
  specific codes are used for measures related to the guideline recommendations for grade of advice for insufficient physical activity, unhealthy eating habits, hazardous use of alcohol and tobacco use and prescribed physical activity
Change in S-NoMAD score (Swedish translation of NoMAD | Change from baseline S-Nomad score up to 4 to 6 months after end of study completion
  23-item questionnaire covering the constructs coherence, cognitive participation, collective action and reflexive monitoring
Change in S-NoMAD score (Swedish translation of NoMAD | Change from baseline S-Nomad score up to 16 to 18 months after end of study completion
  23-item questionnaire covering the constructs coherence, cognitive participation, collective action and reflexive monitoring

SECONDARY OUTCOMES:
Change in perceived clincial intervention by a study specific questionnaire | Change from baseline up to 4 to 6 months after end of implementation support
  Questions related to the patients' perception on receiving the clinical intervention or not
Change in perceived appropriateness (AIM), feasability (FIM) and acceptability (IAM) of the clinical intevention. | Change from baseline in AIM,IAM and FIM up to 4 to 6 months after end of implementation support
  Appropriateness, feasability, acceptability of the clinical intervention is rated on a 5-graded scale with 4 items per construct
Change in perceived appropriateness (AIM), feasability (FIM) and acceptability (IAM) of the clinical intevention. | Change from baseline in AIM,IAM and FIM up to 16 to18 months after end of implementation support
  Appropriateness, feasability, acceptability of the clinical intervention is rated on a 5-graded scale with 4 items per construct

OTHER OUTCOMES:
Interviews to tailor strategies and evaluate implementation process | Interviews pre-intervention and up to 3 to 6 months after end of implementation support
  Semi-structured interview guides directed to facilitators, co-workers and managers
Interviews to evaluate implementation support, clinical process and thoughts about up-scaling | Interviews pre-intervention and up to 16 to18 months after end of implementation support
  Semi-structured interview guides directed to facilitators, co-workers and managers
Person centered processmapping | At baseline
  Structured workshop with patient representatives
Study specific logbook | Through study completion, in average 16 months
  To measure fidelity, dose and reach and changes at the unit that may affect the implementation process

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Nilsagård, Study Director — University Health Care Research Center, Region Örebro County
Locations (1):
- Region Örebro County, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
We don't collect individual data other than in the qualitative parts and we don't have ethical approval to share that

REFERENCES:
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Wandell PE, de Waard AM, Holzmann MJ, Gornitzki C, Lionis C, de Wit N, Sondergaard J, Sonderlund AL, Kral N, Seifert B, Korevaar JC, Schellevis FG, Carlsson AC. Barriers and facilitators among health professionals in primary care to prevention of cardiometabolic diseases: A systematic review. Fam Pract. 2018 Jul 23;35(4):383-398. doi: 10.1093/fampra/cmx137. PMID 29385438
- [Background] Nilsen P, Schildmeijer K, Ericsson C, Seing I, Birken S. Implementation of change in health care in Sweden: a qualitative study of professionals' change responses. Implement Sci. 2019 May 14;14(1):51. doi: 10.1186/s13012-019-0902-6. PMID 31088483
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Elf M, Nordmark S, Lyhagen J, Lindberg I, Finch T, Aberg AC. The Swedish version of the Normalization Process Theory Measure S-NoMAD: translation, adaptation, and pilot testing. Implement Sci. 2018 Dec 4;13(1):146. doi: 10.1186/s13012-018-0835-5. PMID 30509289
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Derived] Nilsagard YE, Smith DR, Soderqvist F, Strid EN, Wallin L. Achieving health-promotion practice in primary care using a multifaceted implementation strategy: a non-randomized parallel group study. Implement Sci Commun. 2025 Apr 7;6(1):36. doi: 10.1186/s43058-025-00723-y. PMID 40197376
- [Derived] Nilsing Strid E, Wallin L, Nilsagard Y. Exploring expectations and readiness for healthy lifestyle promotion in Swedish primary health care: a qualitative analysis of managers, facilitators, and professionals. Scand J Prim Health Care. 2024 Mar;42(1):201-213. doi: 10.1080/02813432.2023.2301556. Epub 2024 Feb 7. PMID 38241166
- [Derived] Strid EN, Wallin L, Nilsagard Y. Expectations on implementation of a health promotion practice using individually targeted lifestyle interventions in primary health care: a qualitative study. BMC Prim Care. 2023 Jun 16;24(1):122. doi: 10.1186/s12875-023-02079-5. PMID 37328813
- [Derived] Strid EN, Wallin L, Nilsagard Y. Implementation of a Health Promotion Practice Using Individually Targeted Lifestyle Interventions in Primary Health Care: Protocol for the "Act in Time" Mixed Methods Process Evaluation Study. JMIR Res Protoc. 2022 Aug 19;11(8):e37634. doi: 10.2196/37634. PMID 35984700

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04799860/Prot_SAP_000.pdf